CLINICAL TRIAL: NCT04685564
Title: A Randomized, Double-blind, Placebo-controlled, Single Dose-escalation, Phase Ia Clinical Study to Evaluate the Safety and Pharmacokinetics of RBD1016 in Healthy Subjects
Brief Title: A Single Dose-escalation Study to Evaluate the Safety and Pharmacokinetics of RBD1016
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Ribo Life Science Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RBHB1101-A
Record Dates: First submitted 2020-12-08; First posted 2020-12-28 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RBD1016 experiment group (Experimental): Subjects in experiment groups will receive a single subcutaneous injection of RBD1016.
  Interventions: Drug: RBD1016
- placebo gruop (Placebo Comparator): Subjects in placebo groups will receive a single subcutaneous injection of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RBD1016 — "Sentinel cohort" design is used in each cohort: each cohort will be administered in two batches, the first 2 subjects will receive RBD1016 or placebo respectively, and safety assessment will be done on D8±1. After safety is confirmed through SRC assessment, the remaining 6 subjects will be randomly assigned to receive RBD1016 or placebo in a ratio of 5:1. SRC will assess the safety after all the subjects in each cohort complete the 28-day safety observation and the subjects may proceed to the next dose cohort with permission.
  Only after all the subjects in the previous dose cohort have completed the safety assessment by SRC (observed for 28 days) may the next dose cohort be initiated with permission.
  Arms: RBD1016 experiment group
Drug: Placebo — the same as RBD1016
  Arms: placebo gruop

SUMMARY:
This is a single dose-escalation phase Ⅰa clinical study to observe the safety and pharmacokinetic profiles of RBD1016 in healthy subjects.

The study consists of screening period (Day -28 to Day -1), treatment period (Day 1 to Day 2), safety assessment period (to Day 29) and safety follow-up period (up to Day 85).

DETAILED DESCRIPTION:
It is a randomized, double-blind, placebo-controlled, single dose-escalation, phase Ia study. The study will enroll 40 healthy subjects, including 5 dose escalation cohorts for dose escalation with 0.3 mg/kg body weight as the starting dose.

After a single-dose injection, there will be a 4-week safety assessment and monitoring phase (Days 1-29). Blood samples for PK analysis will be collected within 60 minutes before dosing, and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h after dosing, respectively. According to the previous PK results, the subsequent PK blood collection points can be adjusted. Total urine samples will be collected once before dosing and in each of 2 time periods after dosing: 0~8 h and 8~24 h. The total urine output will be recorded, and some urine samples will be collected in each time period to analyze and detect the urine drug concentration.

Subjects will undergo safety follow-up from Day 29 to Day 85.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily participate in this clinical trial, are able to correctly understand and have signed the informed consent in writing;
2. Male or female volunteers aged between 18 and 45 years (inclusive);
3. Body weight: male ≥ 50 kg, female ≥ 45 kg; Body Mass Index (BMI) of 18-30 kg/m2 (inclusive);
4. Vital signs, physical examination, 12-lead ECG, and clinical laboratory tests results are within normal range or beyond the normal range but are not clinically significant at the discretion of the investigator.
5. Subjects who are able to use effective methods of contraception throughout the study and within 6 months after the last administration of the investigational product (refer to Appendix 3 for details);
6. Subjects who are able to cooperate with the investigator, comply with study requirements and complete the study in accordance with relevant procedures of the protocol.

Exclusion Criteria:

1. Subjects with positive hepatitis B surface antigen (HBsAg), HCV antibody or HIV antibody; or subjects with concomitant drug-induced or autoimmune hepatopathy (e.g. positive antinuclear antibody [ANA])
2. Medical history of organ transplant or malignancy.
3. Subjects with clinically significant allergic disease or allergic predisposition or with clear allergy to this product or its composition.
4. Subjects with a history of any serious clinical disease or with clear circulatory system, endocrine system, central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system, immune system or metabolic disorder, or with other diseases inappropriate for entry into this study (e.g. history of psychosis), which are clinically significant at the discretion of the investigator.
5. Creatinine clearance (Ccr) <60ml/min [calculation formula: Ccr: (140-age)×body weight (kg)/0.818×Scr (μmol/L), female ×0.85].
6. History of immune-mediated disease (such as: primary thrombocytopaenic purpura, systemic lupus erythematosis, rheumatoid arthritis, autoimmune hemolytic anemia, serious psoriasis, or any other autoimmune disease) which is clinically significant at the discretion of the investigator.
7. Subjects with acute infection (e.g. influenza) in recent 2 weeks.
8. Subjects who have participated in another clinical study and have received another investigational drug within 1 months before treatment initiation.
9. Subjects with other factors which are unsuitable for study participation at the discretion of the investigators.

NOTE: additional inclusion/exclusion criteria may apply, per protocol

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety assessment, AE and SAE of ascending single dose of RBD1016 in healthy subjects. | up to Day 29
  Incidence, nature, and severity of adverse events (AEs) and serious adverse events (SAEs) will be assessed by CTCAE v5.0.
To evaluate the safety assessment, 12-lead ECG of ascending single dose of RBD1016 in healthy subjects. | up to Day 29
  The corrected QT (QTcB) value(ms) from baseline will be reviewed by 12-lead electrocardiogram (12-lead ECG).Data from 12-lead ECG will be summarized descriptively by visit, and flagged abnormalities will be listed.
To evaluate the safety assessment, vital signs of ascending single dose of RBD1016 in healthy subjects. | up to Day 29
  Vital signs includes systolic blood pressure(mm Hg), diastolic blood pressure(mm Hg), pulse rate(beats per minute), body temperature(℃), respiration(beats per minute).Data from vital signs will be summarized descriptively by visit, and flagged abnormalities will be listed.
To evaluate the safety assessment, physical examinations of ascending single dose of RBD1016 in healthy subjects. | up to Day 29
  Physical examinations include weight(kg) and height(m), skin and mucosa, lymph nodes, head and neck, chest, abdomen, spine and limbs, musculoskeletal system, and nervous system. Weight and height will be combined to report BMI in kg/m^2 and other examination results of each area shall be recorded as normal or abnormal. Any abnormalities should be explained in detail, and persistent abnormalities should be recorded at each visit.
To evaluate the safety assessment, clinical lab examinations of ascending single dose of RBD1016 in healthy subjects. | up to Day 29
  Clinical lab examinations, including hematology, urinalysis, biochemistry and coagulation tests.Clinical lab examinations' data in each group will be summarized by listing the categorical changes and summary statistics of source data as well as the change from baseline at each visit (mean, median, standard deviation, range).

SECONDARY OUTCOMES:
To characterize the pharmacokinetic parameter Cmax of RBD1016 in healthy subjects. | within 60 minutes before dosing, and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours after dosing
  Maximum concentration (Cmax)
To characterize the pharmacokinetic parameter AUC0-t of RBD1016 in healthy subjects. | within 60 minutes before dosing, and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours after dosing
  Area under the concentration-time curve from 0 to the collection time t (AUC0-t)
To characterize the pharmacokinetic paramete AUC0-inf of RBD1016 in healthy subjects. | within 60 minutes before dosing, and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours after dosing
  Area under the concentration-time curve from 0 to infinity (inf) (AUC0-inf)
To characterize the pharmacokinetic paramete Tmax of RBD1016 in healthy subjects. | within 60 minutes before dosing, and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours after dosing
  Time to maximum concentration (Tmax)
To characterize the pharmacokinetic paramete t1/2 of RBD1016 in healthy subjects. | within 60 minutes before dosing, and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours after dosing
  Plasma Half-Life (t1/2)
To characterize the pharmacokinetic paramete Vz/F of RBD1016 in healthy subjects. | within 60 minutes before dosing, and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours after dosing
  Volume of distribution in the terminal elimination period (Vz/F)
To characterize the pharmacokinetic paramete λz of RBD1016 in healthy subjects. | within 60 minutes before dosing, and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours after dosing
  Terminal rate constant (λz)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Dr. Lemech, Principal Investigator — Scientia Clinical Research Ltd.
Locations (1):
- Scientia Clinical Research Ltd, Randwick, Australia